CLINICAL TRIAL: NCT01218191
Title: Acute Neurocardiogenic Injury After Subarachnoid Hemorrhage Assessed With Cardiac 18F-FDG PET and 123I-MIBG Scintigraphy: a Prospective Observational Study.
Brief Title: Acute Neurocardiogenic Injury After Subarachnoid Hemorrhage.
Acronym: HSA-2
Status: Completed | Type: Observational
Sponsor: Direction Centrale du Service de Santé des Armées (Other)
Responsible Party: Principal Investigator, PRUNET Bertrand, MD,MSc, Direction Centrale du Service de Santé des Armées
Other Study IDs: HSA-2
Record Dates: First submitted 2010-10-06; First posted 2010-10-11 (Estimated); Last update posted 2012-02-20 (Estimated); Status verified 2012-02

CONDITIONS: Subarachnoid Hemorrhage
Keywords: subarachnoid hemorrhage; scintigraphy; neurocardiogenic injury
MeSH Terms: conditions — Subarachnoid Hemorrhage

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Subarachnoid hemorrhage: Patients presenting a SAH

SUMMARY:
The aim of this study is to describe acute neurocardiogenic injury after subarachnoid hemorrhage assessed with cardiac 123I-MIBG scintigraphy and 18F-FDG PET/CT during the first week and the first six months after SAH.

The study hypothesis is that the evolution of the cardiac disturbances follows the clinical evolution.

DETAILED DESCRIPTION:
The cardiac metabolic disturbance are assessed by a 18F-FDG PET/CT in the first week after SAH and monthly until normal result.

The myocardial sympathetic innervation is assessed by a cardiac 123I-MIBG scintigraphy in the first week after SAH and six months later.

Clinical outcome is assessed by Glasgow Outcome Scale, modified Rankin Scale and MOS-SF36 at 1, 3 and 6 months after SAH.

ELIGIBILITY:
Inclusion Criteria:

* age
* SAH
* Hospitalization in the Military Teaching Hospital Sainte Anne

Exclusion Criteria:

* Refusal of consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients presenting a SAH
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2010-02; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
cardiac 18F-FDG PET | first week after SAH

SECONDARY OUTCOMES:
cardiac 123I-MIBG scintigraphy | first week after SAH
cardiac 18F-FDG PET | one month after first cardiac 18F-FDG PET
cardiac 123I-MIBG scintigraphy | Six months after SAH

CONTACTS AND LOCATIONS:
Overall Officials: Eric MEAUDRE, Professor, Study Director — Military Teaching Hospital Sainte Anne
Locations (1):
- Intensive Care Unit, Military Teaching Hospital sainte Anne, Toulon, France

REFERENCES:
- [Background] Banki NM, Kopelnik A, Dae MW, Miss J, Tung P, Lawton MT, Drew BJ, Foster E, Smith W, Parmley WW, Zaroff JG. Acute neurocardiogenic injury after subarachnoid hemorrhage. Circulation. 2005 Nov 22;112(21):3314-9. doi: 10.1161/CIRCULATIONAHA.105.558239. Epub 2005 Nov 14. PMID 16286583
- [Result] Meaudre E, Jego C, Kenane N, Montcriol A, Boret H, Goutorbe P, Habib G, Palmier B. B-type natriuretic peptide release and left ventricular filling pressure assessed by echocardiographic study after subarachnoid hemorrhage: a prospective study in non-cardiac patients. Crit Care. 2009;13(3):R76. doi: 10.1186/cc7891. Epub 2009 May 20. PMID 19454040
- [Derived] Prunet B, Basely M, D'Aranda E, Cambefort P, Pons F, Cimarelli S, Dagain A, Desse N, Veyrieres JB, Jego C, Lacroix G, Esnault P, Boret H, Goutorbe P, Bussy E, Habib G, Meaudre E. Impairment of cardiac metabolism and sympathetic innervation after aneurysmal subarachnoid hemorrhage: a nuclear medicine imaging study. Crit Care. 2014 Jun 25;18(3):R131. doi: 10.1186/cc13943. PMID 24964817